CLINICAL TRIAL: NCT04752319
Title: BreEStim for Post-Stroke Motor Recovery
Brief Title: BreEStim for Motor Recovery in Chronic Stroke With Moderate Impairment After a Long-term Use (Pilot).
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Sheng Li, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-20-1286 (Experiment 3)
Record Dates: First submitted 2021-02-10; First posted 2021-02-12 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Motor Recovery
Keywords: Finger flexor spasticity; Motor Recovery; BreEStim

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- BreEStim (Experimental): BreEStim is voluntary breathing controlled transcutaneous electrical nerve stimulation.
  Interventions: Device: BreEStim
- EStim (Experimental): EStim is transcutaneous electrical nerve stimulation.
  Interventions: Device: EStim

INTERVENTIONS:
Device: BreEStim — BreEStim will be applied for 10 to 20 minutes per session for multiple sessions
  Arms: BreEStim
Device: EStim — EStim will be applied for 10 to 20 minutes per session for multiple sessions
  Arms: EStim

SUMMARY:
The overall goal is to investigate the effectiveness of a novel intervention - Breathing-controlled electrical stimulation (BreEStim) on finger flexor spasticity reduction and hand function improvement in chronic stroke with moderate impairment after a long-term use.

ELIGIBILITY:
Inclusion criteria:

* has post stroke ≥ 6 months , medically stable;
* Unilateral, single stroke (no restriction on type (ischemic or hemorrhagic) or volume (large or small) of stroke);
* MAS score ≥ 1, i.e., detectable finger flexor hypertonia;

Exclusion criteria include:

* Patients with visual deficit/neglect; hearing or cognitive impairment;
* Patients with history of pulmonary disease (Asthma, chronic obstruction pulmonary disease, COPD);
* Patients that are currently adjusting tone alternating medications (e.g., baclofen), or
* Patients received botulinum toxin injection to the arm/fingers <4 months, or phenol injections < 2 years;
* Patients with a pacemaker;
* Women who are pregnant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in finger flexor spasticity measured by Modified Ashworth Scale (MAS) | Baseline, after 10 intervention sessions, about 3 weeks
  MAS will be performed to check changes of finger flexor spasticity after one session of treatment.
  The Modified Ashworth scale (MAS) scoring is categorical and ranges from 0 to 4, as follows:
  0: No increase in muscle tone
  1. Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension 1+: Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the range of motion (ROM)
  2. More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved
  3. Considerable increase in muscle tone, passive movement difficult
  4. Affected part(s) rigid in flexion or extension

SECONDARY OUTCOMES:
Change in finger extensors and hand function measured by Fugl Myer Assessment (FMA) Scale | Baseline, after 10 intervention sessions, about 3 weeks
  FMA will be assessed to test function changes of finger extensors and hand function after one session of treatment.
  The upper limb motor function domain of the FMA scale will be used, and the score range for this domain is 0 to 66, with a higher score indicating better function.

CONTACTS AND LOCATIONS:
Overall Officials: Sheng Li, MD, PhD, Principal Investigator — University of Texas
Locations (1):
- The University of Texas Health Science Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No